CLINICAL TRIAL: NCT02256488
Title: A Phase III, Multicenter, Randomized, Double-Blind, Controlled Study to Evaluate the Safety and Immunogenicity of Two Trivalent Subunit Influenza Vaccines in Healthy Adult Subjects
Brief Title: Safety and Immunogenicity of Two Trivalent Subunit Influenza Vaccines in Healthy Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: V58_23
Record Dates: First submitted 2014-09-26; First posted 2014-10-03 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Prophylaxis: Influenza

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- TIVc-Lot A (Experimental): Subjects 18 to ≤ 49 years of age who received one vaccination with an investigational vaccine TIVc from Lot A
  Interventions: Biological: TIVc_LOT A
- TIVc-Lot B (Experimental): Subjects 18 to ≤ 49 years of age who received one vaccination with an investigational vaccine TIVc from Lot B
  Interventions: Biological: TIVc_LOT B
- TIVc-Lot C (Experimental): Subjects 18 to ≤ 49 years of age who received one vaccination with an investigational vaccine TIVc from Lot C
  Interventions: Biological: TIVc_LOT C
- TIVf (Active Comparator): Subjects 18 to ≤ 49 years of age who received one vaccination of Control vaccine TIVf
  Interventions: Biological: TIVf

INTERVENTIONS:
Biological: TIVc_LOT A — Single IM (Intramuscular) administration dose of 0.5 mL of TIVc
  Arms: TIVc-Lot A
Biological: TIVc_LOT B — Single IM administration dose of 0.5 mL of TIVc
  Arms: TIVc-Lot B
Biological: TIVc_LOT C — Single IM administration dose of 0.5 mL of TIVc
  Arms: TIVc-Lot C
Biological: TIVf — Single IM administration dose of 0.5 mL of TIVf
  Arms: TIVf

SUMMARY:
The purpose of this study is to evaluate the immunologic equivalence of three consecutive lots of a cell based trivalent subunit influenza vaccine (TIVc), and to assess immunogenicity, safety and tolerability of the vaccine and an egg based trivalent subunit influenza vaccine (TIVf).

The study comprised 1 vaccination, 2 clinic visits, 3 reminder calls and 2 blood draws. Female subjects of childbearing potential were tested for pregnancy before the administration of the vaccine and included only if using and agreeing to continue to use contraception during the course of the study.

The total study participation time per subject is about 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 through 49 years of age.
* Subjects having provided informed consent.
* Individuals in good health

Exclusion Criteria:

* Chronic or acute illness that would interfere with the subject's safety and/or could interfere with the evaluation of study vaccine, including known history of anaphylaxis, serious vaccine reactions or hypersensitivity, known immunodeficiency or receiving immunosuppressive therapy.
* Female of childbearing potential not using acceptable contraceptive methods, pregnant or breastfeeding.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1561 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Anaheim Clincial Trials, Anaheim, California
  - Northern California Clinical Research Center, Redding, California
  - Southern California CRC, San Diego, California
  - Broward Research Group, Hollywood, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Palm Bech Research, West Palm Beach, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Johnson County Clin-Trials, LLC, Lenexa, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Milford Emergency Associate,Inc, Milford, Massachusetts
  - Meridian Clinical Research, Omaha, Nebraska
  - Rochester Clinical Research, Inc, Rochester, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Hickory, Hickory, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Columbia Research Group, Inc, Portland, Oregon
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Research Solutions, LLC, Franklin, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Foothill Family Clinc South, J. Lewis Research Inc., Salt Lake City, Utah
  - Foothill Family Clinic, J. Lewis Research Inc., Salt Lake City, Utah
  - Jordan River Family Medicine, J. Lewis Research, Inc., South Jordan, Utah
  - Clinical Research Associates, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Twenty five study centers in the United States of America.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- TIVc_LOT A: Subjects 18 to ≤ 49 years of age who received one vaccination with an investigational vaccine TIVc from Lot A
- TIVc_LOT B: Subjects 18 to ≤ 49 years of age who received one vaccination with an investigational vaccine TIVc from Lot B
- TIVc_LOT C: Subjects 18 to ≤ 49 years of age who received one vaccination with an investigational vaccine TIVc from Lot C
Period: Overall Study
Arm/Group | TIVc_LOT A | TIVc_LOT B | TIVc_LOT C | TIVf
Started | 387 | 392 | 392 | 390
Completed | 379 | 386 | 382 | 384
Not Completed | 8 | 6 | 10 | 6
Not completed — Lost to Follow-up | 6 | 6 | 9 | 3
Not completed — OTHER | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIVc_LOT A | TIVc_LOT B | TIVc_LOT C | TIVf | Total
Number analyzed (Participants) | 387 | 392 | 392 | 390 | 1561
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (9.1) | 33.1 (8.8) | 33.8 (8.8) | 33.2 (9.0) | 33.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 221 | 227 | 243 | 250 | 941
  MALE | 166 | 165 | 149 | 140 | 620

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Equivalence of 3 Consecutive Influenza Vaccine (TIVc) Production Lots.
Description: Hemagglutination inhibition (HI) geometric mean titers (GMTs) achieved by subjects, for each three vaccine strains, three weeks after one vaccination of one lot of TIVc vaccine (Day 22), evaluated using HI antigen assay.
Time Frame: Day 22
Population: Per Protocol Set(PPS) All subjects in the FAS (Full Analysis Set) Immunogenicity Population who were not excluded due to reasons defined prior to unblinding or analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TIVc_LOT A | TIVc_LOT B | TIVc_LOT C
Number analyzed (Participants) | 363 | 375 | 374
Titers
  A/Brisbane/10/2010 (H1N1) | 667 [595 to 747] | 738 [660 to 824] | 655 [586 to 733]
  A/Texas/50/2012 (H3N2) | 466 [417 to 519] | 472 [424 to 525] | 437 [392 to 486]
  B Massachusetts/2/2012 (B) | 178 [161 to 196] | 175 [159 to 192] | 172 [156 to 189]
Statistical Analysis 1: Comparison: TIVc_LOT A vs TIVc_LOT B; To demonstrate immunologic equivalence of three consecutive TIVc production lots as evaluated by HI antibody responses after vaccination for all 3 influenza strains at day 22; Test type: Non-Inferiority or Equivalence — The lot-to-lot consistency was claimed if the 2-sided 95% CIs of all the three pairwise comparisons was within the equivalence ranges, that is: (μlot A - μlot B) > -0.176 and (μlot A - μlot B) < 0.176 and (μlot A - μlot C) > -0.176 and (μlot A - μlot C) < 0.176 and (μlot B - μlot C) > -0.176 and (μlot B - μlot C) < 0.176; ANCOVA; Ratio of GMTs = 0.9, 95% CI 2-sided [0.667 to 1.5]
Statistical Analysis 2: Comparison: TIVc_LOT A vs TIVc_LOT C; To demonstrate immunologic equivalence of three consecutive TIVc production lots as evaluated by HI antibody responses after vaccination for for all 3 influenza strains at day 22; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of GMTs = 1.02, 95% CI 2-sided [0.667 to 1.5]
Statistical Analysis 3: Comparison: TIVc_LOT B vs TIVc_LOT C; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of GMTs = 1.12, 95% CI 2-sided [0.667 to 1.5]

2. Secondary Outcome: Percentages of Subjects Who Achieved HI Seroconversion and HI Titer ≥1:40 Against Each of Three Strains After One Vaccination of TIVc and TIVf Vaccine.
Description: Percentages of subjects achieving HI seroconversion after each of three vaccine strains were measured three weeks after vaccination of TIVc or TIVf vaccine (day 22).
  Percentages of subjects who achieved HI titer ≥1:40 against each of three vaccine strains were measured three weeks after one vaccination of TIVc or TIVf vaccine.
  HI assay analysis for TIVc vaccine was based on cell-based antigen and for TIVf vaccine was based on egg based antigen.
  According to Center for Biologics Evaluation and Research recommendations (CBER 2007), CBER criteria are met when the lower limit of the 2-sided 95% CI for seroconversion/significant increase is ≥ 40%, and the lower limit of the 2-sided 95% CI for HI titers ≥ 1:40 is ≥ 70%.
Time Frame: Day 22
Population: FAS(Full Analysis Set) All subjects in the Enrolled Population who: ▫ receive a study vaccination and provide immunogenicity data at Day 1 and at Day 22 FAS populations was analyzed "as randomized" (i.e., according to the vaccine a subject was designated to receive, which may be different from the vaccine the subject actually received).
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- TIVc (3 TIVc Lots Pooled): Subjects 18 to ≤ 49 years of age who received one vaccination of an investigational vaccine TIVc
Arm/Group | TIVc (3 TIVc Lots Pooled) | TIVf
Number analyzed (Participants) | 1144 | 379
percentages of subjects
  Influenza A H1N1 Brisbane/2010 CC Ab-SC(1143,379 ) | 60 [57 to 62] | 69 [64 to 74]
  A/Texas/50/2012 (H3N2)- Seroconversion | 49 [46 to 52] | 63 [58 to 68]
  B Massachusetts/2/2012 (B) - Seroconversion | 39 [36 to 42] | 45 [40 to 50]
  Influenza A H1N1 Brisbane/2010 CC Ab-HI ≥1:40Day22 | 99 [99 to 100] | 99 [98 to 100]
  A/Texas/50/2012 (H3N2)- HI ≥1:40(Day 22) | 100 [99 to 100] | 100 [99 to 100]
  B Massachusetts/2/2012 (B) - HI ≥1:40 (Day 22) | 98 [97 to 99] | 92 [89 to 95]

3. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Adverse Events After One Vaccination of TIVc and TIVf
Description: Safety was assessed as the number of subjects who reported solicited local and systemic adverse events from day 1 up to and including day 7 after vaccination of TIVc and control vaccines.
Time Frame: Day 1 through day 7 (without 30 min)
Population: Solicited Safety Set-All subjects in the exposed set with any solicited AE data postvaccination or indicators of solicited AEs postvaccination
Measure: Number; unit: Subjects
Groups:
- TIVf: Subjects 18 to ≤ 49 years of age who received one vaccination of Control vaccine TIVf;
Arm/Group | TIVc (3 TIVc Lots Pooled) | TIVf
Number analyzed (Participants) | 1169 | 391
Subjects
  Induration: number analyzed (Participants) | 1166 | 390
  Induration | 168 | 62
  Erythema: number analyzed (Participants) | 1166 | 390
  Erythema | 208 | 77
  Ecchymosis: number analyzed (Participants) | 1166 | 390
  Ecchymosis | 76 | 30
  Pain | 481 | 135
  Nausea | 91 | 30
  Myalgia | 109 | 28
  Arthralgia | 84 | 28
  Headache | 259 | 80
  Fatigue | 221 | 77
  Diarrhea | 85 | 47
  Chills | 45 | 11
  Loss of appetite | 66 | 39
  Vomiting | 18 | 9
  Fever (≥38°C) | 7 | 2

4. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: Safety was assessed as the number of subjects who reported Unsolicited Adverse Events after vaccination of TIVc and control vaccine.
Time Frame: Day 1 through day 22
Population: Unsolicited Safety Set-All subjects in the exposed set with unsolicited AE data postvaccination.
Measure: Number; unit: Subjects
Arm/Group | TIVc (3 TIVc Lots Pooled) | TIVf
Number analyzed (Participants) | 1169 | 391
Subjects
  Any AE | 139 | 38
  Possibly or probably related AE | 50 | 14
  SAE | 0 | 2
  Possibly or probably related SAE | 0 | 1
  AE leading to withdrawal | 0 | 0
  Medically attended AE | 28 | 9
  New Onset of Chronic Disease | 2 | 1
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period, (Day 1 through Day 22)
Description: SAEs were collected from day 1 through day 22. Unsolicited non-SAEs were also collected through day 22.
  1560 of 1561 subjects received study vaccination and were included in the safety analysis. 1 subject was a screen failure and did not receive study vaccination. 1 subject was randomized to TIVc Lot C, received TIVf, and 1 subject was randomized to TIVc Lot B, received TIVc Lot C vaccine. In the safety analysis 1169 subjects were included in TIVc pooled and 391 subjects in TIVf.
Groups:
- TIVc Pooled: Subjects 18 to ≤ 49 years of age who received one vaccination of an investigational vaccine TIVc
- Total: Total number of subjects
Arm/Group | TIVc Pooled | TIVf | Total
Serious Adverse Events (participants affected / at risk) | 0/1169 | 2/391 | 2/1560
Other Adverse Events (participants affected / at risk) | 709/1169 | 237/391 | 946/1560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc Pooled (N=1169) | TIVf (N=391) | Total (N=1560)
APPENDICITIS (Infections and infestations) | 0 | 1 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc Pooled (N=1169) | TIVf (N=391) | Total (N=1560)
DIARRHOEA (Gastrointestinal disorders) | 86 | 47 | 133
NAUSEA (Gastrointestinal disorders) | 91 | 30 | 121
FATIGUE (General disorders) | 222 | 77 | 299
INJECTION SITE ERYTHEMA (General disorders) | 208 | 77 | 285
INJECTION SITE HAEMORRHAGE (General disorders) | 76 | 30 | 106
INJECTION SITE INDURATION (General disorders) | 168 | 62 | 230
INJECTION SITE PAIN (General disorders) | 481 | 135 | 616
DECREASED APPETITE (Metabolism and nutrition disorders) | 66 | 39 | 105
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 84 | 29 | 113
MYALGIA (Musculoskeletal and connective tissue disorders) | 110 | 28 | 138
HEADACHE (Nervous system disorders) | 262 | 82 | 344

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site was postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.